CLINICAL TRIAL: NCT00236392
Title: Double-Blind Placebo-Controlled Randomized Withdrawal Trial Assessing the Efficacy and Tolerability of "On-Demand" Maintenance Therapy With 10mg o.d. Rabeprazole for 6 Months in Non-Erosive Reflux Disease Patients With Complete Symptom Relief After 4 Week Open Acute Phase
Brief Title: A Study of Efficacy and Safety of "On-demand" Maintenance Therapy With Rabeprazole in Patients With Non-erosive Reflux Disease (NERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003121
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Gastroesophageal Reflux; Heartburn
Keywords: Gastroesophageal reflux; Heartburn; Rabeprazole; Anti-ulcer agents; GERD; Proton pump inhibitor; GORD; Non-Erosive Reflux Disease; NERD
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Non-Erosive Reflux Disease | interventions — Rabeprazole

INTERVENTIONS:
Drug: rabeprazole

SUMMARY:
The purpose of this study is to assess the efficacy and safety of long-term, "on-demand" maintenance therapy with rabeprazole in patients with non-erosive reflux disease (NERD).

DETAILED DESCRIPTION:
More than half of patients with typical gastroesophageal reflux symptoms such as heartburn are considered to have non-erosive reflux disease (NERD), which is characterized by a lack of clinically defined damage to the esophagus. One approach to maintain control of these symptoms is to have medication available "on-demand." This is a double-blind, placebo-controlled study of the effectiveness of "on-demand" rabeprazole in the long-term maintenance of heartburn control in NERD patients, for whom heartburn was resolved with short-term, daily rabeprazole therapy. The study has two phases: an acute phase (4 weeks) during which patients receive rabeprazole medication daily, and an "on-demand" phase (6 months) during which patients take medication (rabeprazole or placebo) as needed. Only patients who have complete resolution of heartburn at the end of the acute phase are eligible to continue in the "on-demand" phase. Efficacy assessments include the proportion of patients discontinuing treatment in the "on-demand" phase because of insufficient heartburn control, and the severity of heartburn and patient satisfaction determined at the beginning and end of "on-demand" phase. Safety assessments include incidence of adverse events throughout the study, physical examination at study initiation, and vital signs at the beginning and the end of the study. The study hypothesis is that "on-demand" therapy with rabeprazole is superior to placebo in maintaining heartburn control and is well tolerated by the patients with NERD. Rabeprazole tablet (10 milligrams[mg]) once daily in the morning for 4 weeks. Rabeprazole tablets (10mg) once daily on an "on-demand" basis for the following 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 12 months history of heartburn as the predominant symptom with at least 2 symptomatic episodes
* Negative endoscopy (no erosive lesions according to the Modified Savary-Miller scale) within 7 days prior to acute treatment
* at least 3 days with moderate to very severe heartburn within one week prior to acute treatment

Exclusion Criteria:

* No known gastro-duodenal ulcer
* no infections, inflammations, or obstruction of the small or large intestine
* no history of gastrointestinal cancer, or prior surgery of the stomach or intestine
* no stomach or abdominal pain or discomfort as the predominant symptom or that requires treatment
* no history of erosive reflux causing inflammation of the esophagus
* no stricture of the esophagus, stomach, or any condition that causes difficulty in swallowing
* no history of non-erosive reflux disease (NERD) that is or was refractory to an adequate treatment course (1 month) with proton pump inhibitors
* no females who are pregnant or those lacking adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2001-10; Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients discontinuing treatment in "on-demand" phase (6 months) because of insufficient heartburn control.

SECONDARY OUTCOMES:
Severity and control of heartburn, overall quality of life (Psychological General Well-Being Index), antacid consumption, and patient satisfaction at the beginning and end of the "on-demand" phase. Incidence of adverse events throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.

REFERENCES:
- [Result] Bytzer P, Blum A, De Herdt D, Dubois D; Trial Investigators. Six-month trial of on-demand rabeprazole 10 mg maintains symptom relief in patients with non-erosive reflux disease. Aliment Pharmacol Ther. 2004 Jul 15;20(2):181-8. doi: 10.1111/j.1365-2036.2004.01999.x. PMID 15233698